CLINICAL TRIAL: NCT03547414
Title: Does Urinary TIMP2 and IGFBP7 Can Identify High Risk Patients of Progression From Mild and Moderate to Severe Acute Kidney Injury During Septic Shock? HEMOCHECK
Brief Title: Does Urinary TIMP2 and IGFBP7 Can Identify High Risk Patients of Progression From Mild and Moderate to Severe Acute Kidney Injury During Septic Shock?
Acronym: HEMOCHECK
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Centre Hospitalier Universitaire, Amiens (Other)
Responsible Party: Sponsor
Other Study IDs: PI2018_843_0030
Record Dates: First submitted 2018-05-17; First posted 2018-06-06 (Actual); Last update posted 2018-06-06 (Actual); Status verified 2018-06

CONDITIONS: Acute Kidney Injury; Septic Shock
MeSH Terms: conditions — Acute Kidney Injury; Shock, Septic

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Nephrocheck test — A fresh urine sample was collected on inclusion (maximum 6 hours after starting catecholamines) through the urine collecting tube and frozen at -80°C. At the end of the study, urine samples were thawed and centrifuged as recommended by the manufacturer and the urinary TIMP2*IGFBP7 concentration was determined using the Nephrocheck™ test. The Nephrocheck™ test simultaneously measures into the Astute 140™ meter (a bench top analyzer) the urinary concentrations of TIMP2 and IGFBP7 on 100 µl of urine mixed with 100 µl of buffer. The result is expressed as a single number corresponding to the product of TIMP2 and IGFBP7 concentrations.

SUMMARY:
Septic shock is one of the leading causes of death in patients admitted to the intensive care unit (ICU). Acute kidney injury (AKI) occurs in almost 50% of septic patients and is associated with significant mortality. Progression to the last stage (KDIGO stage 3) of AKI is an important step in the disease, as it usually requires initiation of RRT. Renal biomarkers are unable to accurately identify those patients who will progress to severe AKI (KDIGO 3). However, identification of patients at risk of progression to severe AKI could help the clinician to initiate optimal therapy including RRT. A new urine test, the Nephrocheck™ corresponding to the product of the urinary concentrations of 2 markers of renal tubule injury (TIMP2 and IGFBP7) has been validated. The Investigator have already performed two previous studies including septic shock patients (AKICHECK and BIOOCHECK). those previous datas will be reanalysed to examine whether the new urinary biomarkers TIMP2 and IGFBP7 can predict progression within 24 hours and 72 hours from mild and moderate (KDIGO 1 or 2) to severe AKI (KDIGO 3) in patients with septic shock.

-All the datas required will be collected from two previous studies (AKICHECK and BIOCHECK) performed in 3 centers: Amiens medical ICU, Melun medico surgical ICU and Montpellier Medical ICU.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 or over
* Septic shock (according to Bone's criteria) within 4 hours of introduction of catecholamines
* AKI, characterized by a KDIGO score ≥ 1
* Social security coverage

Exclusion Criteria:

* AKI requiring emergency RRT (in the critical care physician's opinion).
* Anuria
* Stage 4-5 chronic kidney failure with a GFR below 30 ml/min.
* Rapidly progressing renal disorders (glomerulonephritis, HUS, blockage, etc.)
* Obstructive AKI
* Probable glomerular damage (nephritic syndrome, nephrotic syndrome, chronic glomerulonephritis)
* Pregnancy or breastfeeding
* Legal guardianship or lack of social security coverage.
* Cardiocirculatory arrest
* Life expectancy <48 hours.
* Child C cirrhosis
* Prior occurrence of AKI during the current hospital stay
* Transplantation
* Subject participating in another study with an exclusion period ongoing at the time of the pre-inclusion

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients with Septic shock (according to Bone's criteria) within 6 hours of introduction of catecholamines
Sampling Method: Non-Probability Sample
Enrollment: 110 (Estimated)
Dates: Start 2018-08-16 (Estimated); Primary Completion 2018-09-16 (Estimated); Study Completion 2018-12-30 (Estimated)

PRIMARY OUTCOMES:
KDIGO classification | 72 hours
  predictive value of Nephrocheck™ with regard to the worsening of AKI, defined as severe AKI (KDIGO 3) in 72 hours following inclusion

REFERENCES:
- [Derived] Maizel J, Daubin D, Vong LV, Titeca-Beauport D, Wetzstein M, Kontar L, Slama M, Klouche K, Vinsonneau C. Urinary TIMP2 and IGFBP7 Identifies High Risk Patients of Short-Term Progression from Mild and Moderate to Severe Acute Kidney Injury during Septic Shock: A Prospective Cohort Study. Dis Markers. 2019 Apr 1;2019:3471215. doi: 10.1155/2019/3471215. eCollection 2019. PMID 31061681